CLINICAL TRIAL: NCT02872285
Title: A Randomized, Placebo-Controlled, Double-Blind Study to Assess the Efficacy and Safety of LYC-30937-EC in Subjects With Moderate Chronic Plaque-Type Psoriasis
Brief Title: An Efficacy and Safety Study of LYC-30937-EC in Subjects With Moderate Chronic Plaque-type Psoriasis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Lycera Corp. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: LYC-30937-2003
Record Dates: First submitted 2016-08-16; First posted 2016-08-19 (Estimated); Results first posted 2019-04-02 (Actual); Last update posted 2019-04-10 (Actual); Status verified 2019-04

CONDITIONS: Psoriasis
MeSH Terms: conditions — Psoriasis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- LYC-30937-EC 25 mg PO once daily (QD) (Experimental): LYC-30937-EC 25 mg by mouth once daily for 12 weeks
  Interventions: Drug: Drug: LYC-30937-EC
- Matching Placebo PO QD (Placebo Comparator): Placebo enteric coated (EC) by mouth once daily for 12 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Drug: LYC-30937-EC
  Arms: LYC-30937-EC 25 mg PO once daily (QD)
Drug: Placebo
  Arms: Matching Placebo PO QD

SUMMARY:
The objective of this Phase 2 trial is to determine the efficacy and safety of LYC-30937-EC in patients with moderate plaque-type psoriasis.

DETAILED DESCRIPTION:
Approximately 30 subjects will be enrolled in this double-blind, placebo-controlled study. The randomization will be stratified 2:1 into the LYC-30937-EC cohort (2) or the placebo cohort (1). The active cohort will receive LYC-30937-EC 25 mg once daily, which demonstrated safety and tolerability in Phase I trials.

The study is designed for patients with previously diagnosed moderate chronic plaque-type psoriasis and consists of the following:

* Screening period (initials assessment and eligibility scoring)
* Day 1: confirm eligibility, baseline efficacy assessments (PASI, IGA), randomize and initiate dosing
* Week 2: safety assessments including vital signs, body temperature, physical exam, clinical labs will be performed
* Week 4: efficacy (PASI, IGA) and safety assessments including vital signs, body temperature, physical exam, and clinical labs will be performed
* Week 8: efficacy (PASI, IGA) and safety assessments including vital signs, body temperature, physical exam, and clinical labs will be performed
* Week 12: final efficacy assessments (PASI, IGA), safety assessments including vital signs, body temperature, physical exam, ECG, and clinical labs will be performed
* Week 14: final safety assessments including vital signs, body temperature, and clinical labs

ELIGIBILITY:
Inclusion Criteria:

* Have a diagnosis of plaque-type psoriasis for at least 6 months prior to screening.
* Must have chronic moderate plaque-type psoriasis confirmed at both screening and baseline visits. Moderate plaque-type psoriasis is defined as a PASI > 7, with body surface area (BSA) involvement 5-15% inclusive and overall lesion severity of "moderate" or "marked, " where "moderate" = plaque elevation (0.75mm), moderate red coloration, coarse scale predominates; "marked" = moderate plaque elevation (1.0mm), bright red coloration, and thick, non-tenacious scale predominates.
* Female subjects of childbearing potential must agree to use two highly effective forms of contraception during study participation and for 30 days after their last dose of treatment of study drug treatment.
* Male subjects with partners of childbearing potential must take appropriate precautions to avoid fathering a child while participating in the study and use appropriate barrier contraception or abstinence during the study and for 30 days after their last dose of study drug.
* Agree to avoid prolonged sun exposure and avoid tanning booths or ultraviolet (UV) light sources during the study.
* Ability to provide written informed consent and to be compliant with the schedule of events.

Exclusion Criteria:

* Non-plaque-type psoriasis (eg, pustular, erythrodermic, and guttate psoriasis).
* Drug-induced psoriasis (ie, new onset or current exacerbation from beta-blockers, calcium channel blockers, or lithium).
* Spontaneously improving or rapidly deteriorating plaque psoriasis.
* Comorbid psoriatic arthritis that is not amenable to treatment with NSAIDs.
* Treatment with a biologic agent for psoriasis.
* Failed 2 or more systemic treatments for plaque psoriasis.
* Received phototherapy or prolonged sun exposure or use of tanning booth or other ultraviolet light source within 4 weeks of initiating screening procedures.
* Received systemic drug therapy (non-biologic) for plaque psoriasis or any systemic medication that could affect psoriasis or its evaluation (PASI or IGA), including but not limited to oral or injectable corticosteroids, retinoids, sulfasalazine, within 4 weeks of initiating screening procedures.
* Received topical medication that could affect psoriasis or its evaluation (PASI or IGA), including but not limited to corticosteroids, retinoids, topical vitamin D derivatives, pimecrolimus, tacrolimus, calcipotriene, within 2 weeks of initiating screening procedures.
* Received immunosuppressant agents (eg, cyclosporine, azathioprine, methotrexate) within 8 weeks of initiating screening procedures.
* Any of the following laboratory abnormalities:

  1. liver function tests > 1.5 x the upper limit of normal (ULN) or direct bilirubin > 1.5 x ULN
  2. hemoglobin < 8.5 g/dl (international system units [SI]: < 85 g/L)
  3. neutrophils < 1500/mm3 (SI: < 1.5 x 109/L)
  4. white blood cell (WBC) count < 3,000/mm3 (SI: < 3.0 x 109/L)
  5. platelets < 80,000 mm3 (SI: 80 x 109/L)
  6. international normalized ratio (INR) > 1.5
  7. serum creatinine > 1.4 mg/dL for women or > 1.6 mg/dL for men
* Clinically relevant hepatic, neurological, pulmonary, dermatological, ophthalmological, gastrointestinal, endocrine, psychiatric, or other major systemic disease making implementation of the protocol or interpretation of the study difficult or that would put the subject at risk by participating in the study.
* History of or currently active primary or secondary immunodeficiency.
* Treatment with an investigational agent within 30 days prior to initiating screening procedures.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2016-12-05 (Actual); Primary Completion 2017-06-22 (Actual); Study Completion 2017-06-22 (Actual)

CONTACTS AND LOCATIONS:
Locations (7):
- United States (7):
  - Lycera Investigational Site, Carmel, Indiana
  - Lycera Investigational Site, Andover, Massachusetts
  - Lycera Investigational Site, Fridley, Minnesota
  - Lycera Investigational Site, East Windsor, New Jersey
  - Lycera Investigational Site, High Point, North Carolina
  - Lycera Investigational Site, Broomall, Pennsylvania
  - Lycera Investigational Site, Norfolk, Virginia

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at 7 study centers within the United States. Study centers were dermatology medical clinics experienced in conducting clinical trials.
Pre-assignment Details: Participants were 18 to 75 years of age with chronic plaque-type psoriasis for ≥ 6 months prior to screening. Eligible patients had a baseline Psoriasis Area and Severity Index (PASI) score > 7 with body surface area (BSA) involvement of 5-15% and overall lesion severity rated as moderate or marked.
Groups:
- LYC-30937-EC 25 mg PO QD: LYC-30937-EC 25 mg by mouth once daily for 12 weeks
  Drug: LYC-30937-EC
- Matching Placebo PO QD: Placebo enteric coated (EC) by mouth once daily for 12 weeks
  Placebo
Period: Overall Study
Arm/Group | LYC-30937-EC 25 mg PO QD | Matching Placebo PO QD
Started | 22 | 11
Completed | 17 | 9
Not Completed | 5 | 2
Not completed — Withdrawal by Subject | 2 | 0
Not completed — Lost to Follow-up | 2 | 2
Not completed — Discontinued due to back surgery | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | LYC-30937-EC 25 mg PO QD | Matching Placebo PO QD | Total
Number analyzed (Participants) | 22 | 11 | 33
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.6 (13.91) | 48.5 (12.96) | 50.6 (13.48)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 5 | 14
  Male | 13 | 6 | 19
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 2
  Not Hispanic or Latino | 21 | 10 | 31
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 0 | 2
  White | 20 | 11 | 31
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Baseline Psoriasis Area and Severity Index (PASI) score [Mean (Standard Deviation); unit: units on a scale] — The PASI is a measure of chronic plaque-type psoriasis disease. It combines lesion severity (erythema, thickness, scaling) and skin surface area involvement in 4 defined anatomical body regions (head, upper extremities, trunk, lower extremities). PASI scores range from 0 to 72 with higher scores indicative of greater disease severity. Lesion severity (erythema, thickness, scaling) is scored on a scale of 0 (none) to 4 (very severe) on each of the 4 body regions. Degree of skin area involvement in each body region is scored on a scale of 0 (no involvement) to 6 (90-100% involvement).
  units on a scale | 9.72 (2.12) | 9.38 (2.66) | 9.61 (2.28)

OUTCOME MEASURES:

1. Primary Outcome: The Mean Percent Change From Baseline to Week 12 in Psoriasis Area and Severity Index (PASI).
Description: This endpoint was calculated in each treatment group by taking the Week 12 PASI score and subtracting the baseline PASI and dividing by the baseline PASI, then multiplying by 100 to get the percent change from baseline. The PASI is a measure of chronic plaque-type psoriasis disease. It combines lesion severity (erythema, thickness, scaling) and skin surface area involvement in 4 defined anatomical body regions (head, upper extremities, trunk, lower extremities). PASI score ranges from 0 to 72 with higher scores indicative of greater disease severity. Lesion severity (erythema, thickness, scaling) is scored on a scale of 0 (none) to 4 (very severe) on each of the 4 body regions. Degree of skin area involvement in each body region is scored on a scale of 0 (no involvement) to 6 (90-100% involvement).
Time Frame: Baseline to Week 12
Population: The full analysis set included all randomized subjects. Randomized subjects included in this analysis had to have both a baseline and a Week 12 PASI score.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | LYC-30937-EC 25 mg PO QD | Matching Placebo PO QD
Number analyzed (Participants) | 18 | 9
percent change | -25.08 (26.43) | -12.63 (19.67)
Statistical Analysis 1: Comparison: LYC-30937-EC 25 mg PO QD vs Matching Placebo PO QD; Subjects included in this analysis had to have both a baseline and Week 12 PASI scores; Test type: Superiority; p = 0.2205, ANCOVA — ANCOVA was used to compare mean percent change in PASI score between baseline and Week 12 between LYC-30937 and placebo treatment groups with treatment as a factor and baseline as a covariate; Mean Difference (Final Values) = -12.80, 95% CI 2-sided [-33.793 to 8.199]

2. Secondary Outcome: The Number of Subjects Who Achieve a ≥ 75% Reduction From Baseline in PASI at Week 12.
Description: This endpoint calculated the number of subjects achieving a ≥ 75% reduction in their Week 12 PASI score compared to their baseline PASI.
  The PASI is a measure of chronic plaque-type psoriasis disease. It combines lesion severity (erythema, thickness, scaling) and skin surface area involvement in 4 defined anatomical body regions (head, upper extremities, trunk, lower extremities). PASI score ranges from 0 to 72 with higher scores indicative of greater disease severity. Lesion severity (erythema, thickness, scaling) is scored on a scale of 0 (none) to 4 (very severe) on each of the 4 body regions. Degree of skin area involvement in each body region is scored on a scale of 0 (no involvement) to 6 (90-100% involvement).
Time Frame: Baseline to Week 12
Population: The full analysis set included all randomized subjects. Randomized subjects included in this analysis were those with PASI scores at baseline and at Week 12.
Measure: Count of Participants; unit: Participants
Arm/Group | LYC-30937-EC 25 mg PO QD | Matching Placebo PO QD
Number analyzed (Participants) | 18 | 9
Participants | 1 | 0
Statistical Analysis 1: Comparison: LYC-30937-EC 25 mg PO QD vs Matching Placebo PO QD; Test type: Superiority; p = 0.4712, Chi-squared; 2-sided p-value

3. Secondary Outcome: The Mean Percent Change From Baseline to Week 12 in Percent Body Surface Area (BSA).
Description: Mean percent change from baseline to Week 12 in %BSA was calculated by taking the Week 12 %BSA and subtracting the baseline %BSA then dividing by the baseline %BSA and multiplying by 100. The mean percent change from baseline to Week 12 in each treatment group were compared using analysis of covariance with treatment as a factor and baseline as a covariate.
Time Frame: Baseline to Week 12
Population: The full analysis set included all randomized subjects. Randomized subjects included in this analysis had to have both a baseline and a Week 12 %BSA score.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | LYC-30937-EC 25 mg PO QD | Matching Placebo PO QD
Number analyzed (Participants) | 18 | 9
percent change | -12.69 (26.18) | -7.68 (35.75)
Statistical Analysis 1: Comparison: LYC-30937-EC 25 mg PO QD vs Matching Placebo PO QD; Test type: Superiority; p = 0.6695, ANCOVA; Mean Difference (Final Values) = -5.34, 95% CI 2-sided [-30.87 to 20.18]

4. Secondary Outcome: The Number of Subjects Who Achieve "Cleared" (Score = 0) or "Minimal" (Score = 1) on the Static Investigators Global Assessment at Week 12.
Description: This endpoint is number of subjects who achieved a score of 0 or 1 on the static IGA at week 12. The static IGA is used to measure psoriasis severity. The static IGA used in this study was a 6-point scale: 0 = Cleared [no plaque elevation, erythema or scaling, hyperpigmentation may be present]; 1 = Minimal [minimal plaque elevation (=0.25mm), faint erythema, minimal scaling with occasional fine scale over < 5% of lesion]; 2 = Mild [mild plaque elevation (=0.5mm), light red coloration, fine scale predominates]; 3 = Moderate [moderate plaque elevation (=0.75mm), moderate red coloration, coarse scale predominates]; 4 = Marked (marked plaque elevation (=1mm), bright red coloration, thick non-tenacious scale predominates]; 5 = Severe (severe plaque elevation (≥1.25mm), dusky to deep red coloration, very thick tenacious scale predominates].
Time Frame: 12 weeks
Population: The full analysis set included all randomized subjects. Randomized subjects included in this analysis had to have both a baseline and a Week 12 static IGA score.
Measure: Count of Participants; unit: Participants
Arm/Group | LYC-30937-EC 25 mg PO QD | Matching Placebo PO QD
Number analyzed (Participants) | 18 | 9
Participants | 1 | 0
Statistical Analysis 1: Comparison: LYC-30937-EC 25 mg PO QD vs Matching Placebo PO QD; Test type: Superiority; p = 0.4712, Chi-squared — 2-sided p-value

5. Secondary Outcome: The Number of Subjects Who Achieve a 2 Step Reduction on the Static Investigators Global Assessment (IGA) at Week 12.
Description: This endpoint is based on number of subjects who achieved a 2 step reduction in the static IGA at week 12 (ie, a score of 5 at baseline to a score of 3 or less at Week 12). The static IGA is used to measure psoriasis severity. The static IGA used in this study was a 6-point scale: 0 = Cleared [no plaque elevation, erythema or scaling, hyperpigmentation may be present]; 1 = Minimal [minimal plaque elevation (=0.25mm), faint erythema, minimal scaling with occasional fine scale over < 5% of lesion]; 2 = Mild [mild plaque elevation (=0.5mm), light red coloration, fine scale predominates]; 3 = Moderate [moderate plaque elevation (=0.75mm), moderate red coloration, coarse scale predominates]; 4 = Marked (marked plaque elevation (=1mm), bright red coloration, thick non-tenacious scale predominates]; 5 = Severe (severe plaque elevation (≥1.25mm), dusky to deep red coloration, very thick tenacious scale predominates].
Time Frame: 12 weeks
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | LYC-30937-EC 25 mg PO QD | Matching Placebo PO QD
Number analyzed (Participants) | 18 | 9
Participants | 1 | 0
Statistical Analysis 1: Comparison: LYC-30937-EC 25 mg PO QD vs Matching Placebo PO QD; Test type: Superiority; p = 0.4712, Chi-squared — 2-sided p-value

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the time subjects signed the study informed consent until the Week 14 follow-up visit. Treatment-emergent adverse events were those adverse events occurring or worsening after the first dose of study drug (LYC-30937-EC or placebo) up to the Week 14 follow-up visit.
Description: AE severity was assessed by the Investigator using the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) v 4.03, with grading as follows: Grade 1 = mild (asymptomatic or mild symptoms), Grade 2 = moderate (minimal, local intervention, or noninvasive intervention indicated); Grade 3 = severe (or medically significant but not life-threatening); Grade 4 = life-threatening; Grade 5 = death.
Arm/Group | LYC-30937-EC 25 mg PO QD | Matching Placebo PO QD
All-Cause Mortality (participants affected / at risk) | 0/22 | 0/11
Serious Adverse Events (participants affected / at risk) | 0/22 | 0/11
Other Adverse Events (participants affected / at risk) | 11/22 | 4/11
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | LYC-30937-EC 25 mg PO QD (N=22) | Matching Placebo PO QD (N=11)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 2 (2) | 0 (0)
Headache (Nervous system disorders) | 2 (6) | 0 (0)
Nasopharyngitis (Infections and infestations) | 2 (2) | 0 (0)
Pruritis (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 2 (2) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (2) | 1 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2)
Fatigue (General disorders) | 0 (0) | 1 (1)
Flatulence (Gastrointestinal disorders) | 0 (0) | 2 (2)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Psoriasis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Seborroea (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Varicose vein (Vascular disorders) | 0 (0) | 1 (1)
Fractured coccyx (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Center results cannot be submitted for publication before results of multicenter study are published unless it is ≥18 months since study completion. Then Investigator can publish if manuscript is submitted to Lycera ≥ 60 days prior to submission (or per Investigator contract). If Lycera decides publication would hinder development, Investigator must delay submission. Investigator must delete confidential information before submission and defer publication to allow patent applications.

DOCUMENTS (2):
  • Study Protocol (2016-08-30): https://cdn.clinicaltrials.gov/large-docs/85/NCT02872285/Prot_000.pdf
  • Statistical Analysis Plan (2017-07-14): https://cdn.clinicaltrials.gov/large-docs/85/NCT02872285/SAP_001.pdf